CLINICAL TRIAL: NCT02380235
Title: Phase IV Clinical Study of Pegylated Somatropin (PEG Somatropin) to Treat Growth Hormone Deficiency Children (Clinical Trial I)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 004 CT-2
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-somatropin (Experimental): 0.12mg/kg/w
  Interventions: Biological: PEG-somatropin
- PEG-Somatropin (Experimental): 0.20mg/kg/w
  Interventions: Biological: PEG-somatropin

INTERVENTIONS:
Biological: PEG-somatropin — 0.20mg/kg/w
Biological: PEG-somatropin — 0.12mg/kg/w

SUMMARY:
This study evaluates the safety and efficiency of Pegylated Somatropin (PEG Somatropin) Injection in the treatment of endogenous growth hormone deficiency (GHD) in the broad of population of children.

ELIGIBILITY:
Inclusion Criteria:

* Before starting treatment, according to the medical history, clinical symptoms and signs, GH stimulation test and imaging examination, patients are diagnosed as GHD.

  * According to the height statistical data of Chinese children's physique development in nine cities in 2005,height is lower than the third percentile of growth curve of normal children with the same age and gender.
  * Height velocity (HV) ≤5.0 cm/yr.
  * GH stimulation test with two different mechanisms affirms that GH peak concentration of patients' plasma<10.0ng/ml.
  * Bone age (BA) ≤9 years in girls and ≤10 years in boys, at least 1 year less than his/her chronological age (CA).
* Be in preadolescence (Tanner stage 1) and have a CA ≧ 3 years.
* Receive no prior GH treatment within 6 months.
* Sign informed consent.

Exclusion Criteria:

* People with abnormal liver or kidney function (ALT> 2 times the upper limit of normal value, Cr> the upper limit of normal value).
* Patients positive for hepatitis B core antigen (HBc), hepatitis B surface antigen (HBsAg) or hepatitis Be antigen (HBeAg).
* People with known highly allergic constitution or allergy to the drug of the study.
* People with severe cardiopulmonary, hematological and malignant tumors diseases or general infection and immune deficiency.
* Diabetic.
* Potential tumor patients (family history).
* Abnormal growth and development, such as Turner syndrome, constitutional delay of growth and puberty,Laron syndrome, growth hormone receptor deficiency, girls of growth retardation without excluding abnormal chromosome.
* Subjects took part in other clinical trial study within 3 months.
* Other conditions which in the opinion of the investigator preclude enrollment into the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Ht SDSca | Baseline, 4,12,26 weeks after initiating treatment
  Ht SDSca was calculated by dividing the difference between the actual height of a patient and the mean height of the population for that chronological age by the standard deviation (SD) of the height of the population for that chronological age

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Children's Hospital Affiliated to Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences &Peking Union Medical College, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital, Jiangnan University, Wuxi, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - West China Second University Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Xin Hua Hospital Affiated to Shanghai Jiao Tong University School of Medicine, Shanghai